CLINICAL TRIAL: NCT00439582
Title: Comparative Effect of 2 Different Sources of Trans Fatty Acid (Milk Fat vs Hydrogenated Oil)on Cardiovascular Risk Factors in Healthy Humans
Brief Title: Trans Fatty Acids and Cardiovascular Risk Factors
Acronym: TRANSFACT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: AU599; 04.28.NRC
Record Dates: First submitted 2007-02-21; First posted 2007-02-23 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2009-03

CONDITIONS: Cardiovascular Disease
Keywords: Lipoproteins; Milk fat; Public health nutrition; trans fatty acid
MeSH Terms: conditions — Cardiovascular Diseases | interventions — polyethoxylated castor oil

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: vaccenic acid enriched milk fat (VAMF) [Transfact1]
- 2 (Experimental)
  Interventions: Dietary Supplement: hydrogenated oil

INTERVENTIONS:
Dietary Supplement: vaccenic acid enriched milk fat (VAMF) [Transfact1]
  Arms: 1
Dietary Supplement: hydrogenated oil — Partially hydrogenated vegetable oils (PHVO) and vegetable oils and fats
  Arms: 2

SUMMARY:
Background:

Detrimental effects of consumption of industrial trans fatty acids (TFA) from partially hydrogenated vegetable oils (PHVO) on cardiovascular disease (CVD) risk factors are well documented. However, very little information is available on the effect of natural sources of TFA coming from milk fat, dairy products and ruminant meat. In fact, due to the naturally low level of TFA in milk fat, it is almost impossible to conduct a clinical trial with a limited number of subjects.

Methodology:

To compare the effects of industrial and natural dietary sources of TFA, two specific test fats have been designed and produced. A substantial amount of milk fat (130 kg) enriched in TFA has been produced by modification of the cow's diet and selection of cows with the highest TFA content. The level obtained was approximately 4- to 7-fold higher than typically present in milk fat ( - 20 instead of 3-6 g/100 g of total fatty acids). The control fat is composed of PHVO balanced in saturated fatty acids (lauric, myristic and palmitic). Both experimental fats contain about 20-22% of monounsaturated TFA and the volunteers' daily experimental fat intake (54 g), will represent about 12.0 g/day of TFA or 5.4% of the daily energy (based on 2000 kcal/day). These two test fats have been incorporated into food items and will be provided to 46 healthy subjects under a randomised, double blind, controlled, cross-over design. The primary outcome is high-density lipoprotein cholesterol (HDL-C), which is an independent risk factor for CVD. Other parameters such as lipoprotein cholesterol (LDL-C), very low-density lipoprotein cholesterol (VLDL-C), and HDL-C level and subclasses will be also to be evaluated.

DETAILED DESCRIPTION:
Design:

This is a double blind, controlled, randomised, cross-over, single center clinical trial.

Product(s) to be tested:

Food items (butter, cheese and biscuits) manufactured using (i) an experimental milk fat and (ii) a mixture of vegetable oils (including partially hydrogenated oils), used as control. Both fats are balanced for their trans fatty acid content and saturated fatty acids content. The main difference of these two experimental fats (milk fat and control fat) is the distribution of trans fatty acids (TFA). The experimental milk fat, entitled "vaccenic acid enriched milk fat" (VAMF), has been obtained by feeding cows with a diet containing sunflower oil. The distribution (the quality) of monounsaturated C18:1 TFA in the VAMF is therefore close to the usual milk fat, but with higher levels (enriched milk).The experimental control fat, shorted CTRL, has been obtained by mixing partially hydrogenated vegetable oils (PHVO) and vegetable oils and fats.

Amount, dosage, route of administration, duration of treatment:

During the 1-week run-in period, subjects should eat daily the same products as the experimental ones (butter, cheese and biscuits) but manufactured using usual milk collected in France. The subjects should then eat daily for 3 weeks butter, cheese and biscuits containing one of the 2 experimental fats (milk fat or control fat, cross-over with 1-week wash-out period) so that they eat daily about 54 g of the experimental fat, which contain about 20-22% of TFA. The total study duration for each subject is 8 weeks: 1-week run-in period, 3-week experimental fat diet in cross-over with 1-week wash-out period between both experimental periods.

All the measurements and blood samplings will be done on the first day of week 1, 3, 4, 5, 7 and 8.

Primary outcome:

HDL-Cholesterol (HDL-C) levels

Secondary outcomes:

* Triglycerides, total cholesterol, Apo A1 , Apo B, factor VII and factor VIIa, fibrinogen levels. Lp(a) and CETP, measured on plasma by fluorimetry. LDL-cholesterol (LDL-C) will be calculated
* LDL, HDL and VLDL levels and subclasses

Other outcome:

evaluation of the fatty acid profiles of plasma cholesteryl esters and phospholipids

ELIGIBILITY:
Inclusion Criteria:

* HDL cholesterol, g/L > 0.4
* Triacylglycerol g/L <1.50
* LDL Cholesterol g/L <1.60
* Affiliated to National Health Insurance
* Waist size < 102 cm (men) or 88 cm (women)
* Normal blood pressure (diastolic <90 mm Hg, systolic <140 mm Hg)
* Normal liver functions (γ-GT, transaminases, alkaline phosphatase)
* Normal white blood cells count (4-10 g/L)
* For women: effective contraception
* Subject giving his/her written informed consent
* Subject willing to comply with the study procedures
* Subject considered as normal after clinical examination and medical questionnaire

Exclusion Criteria:

* Reported food allergies
* Currently participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of this study
* Hepatic or renal impairments
* Positive serologies to HIV or HCV, determined on blood sample
* For women, pregnant or presently attempting to get pregnant (-HCG blood test) or menopause or lactating
* Blood donation done less than 2 months before the start of the study
* Chronic pathologies: diabetes (fasted glycaemia > 6,1 mmol/L), hypertriglyceridemia (≥1.50 g/L), hypertension (systolic blood pressure ≥ 140 mm Hg and/or diastolic blood pressure ≥ 90 mm Hg), cardiovascular diseases, chronic inflammatory diseases
* Intestine, cardiovascular, kidney and cancer pathologies in the last 5 years
* Previous heavy intestine surgery (except appendicectomy)
* Previous medical and/or surgery judged by the investigator as incompatible with this study
* High variation (> 5%) of body weight during the last 3 months
* Consuming nutritional supplements which could interfered with lipid metabolism (fish oil capsule, vitamins, soja lecithins,…)
* Heavy consumer of alcohol (evaluated thanks to the values of the following hepatic enzymes: -GT, ASAT, ALAT)
* Smoker or ex-smoker who stopped smoking less than 1 month before V0
* Practicing intensive physical exercise (> 3 h per week)
* Vegetarian or vegan
* Taking medication for depressive or psychiatric state
* Being under someone's supervision
* Refusal to be registered on the National Volunteers Data file
* Disliking butter, margarine, cheese, biscuits and/or vegetable oil
* Dietary habits unreliable to controlled food intake
* Being in exclusion on the National Volunteers Data file

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46
Dates: Start 2005-08; Study Completion 2005-12

PRIMARY OUTCOMES:
HDL-Cholesterol (HDL-C) levels.

SECONDARY OUTCOMES:
Triglycerides
Total cholesterol
Apo A1
Apo B
Factor VII
Factor VIIa
fibrinogen levels
Lp(a)
LDL, HDL and VLDL levels and subclasses

CONTACTS AND LOCATIONS:
Overall Officials: Yves Boirie, MD, PU-PH, Principal Investigator — UMR1019 INRA - Université Clermont1; Jean-Michel Chardigny, PhD, Study Director — UMR 1019 INRA - Université Clermont1
Locations (1):
- Centre de Recherche en Nutrition Humaine (CRNH), UEN, Laboratoire de Nutrition Humaine, Clermont-Ferrand, France

REFERENCES:
- [Background] Chardigny JM, Malpuech-Brugere C, Dionisi F, Bauman DE, German B, Mensink RP, Combe N, Chaumont P, Barbano DM, Enjalbert F, Bezelgues JB, Cristiani I, Moulin J, Boirie Y, Golay PA, Giuffrida F, Sebedio JL, Destaillats F. Rationale and design of the TRANSFACT project phase I: a study to assess the effect of the two different dietary sources of trans fatty acids on cardiovascular risk factors in humans. Contemp Clin Trials. 2006 Aug;27(4):364-73. doi: 10.1016/j.cct.2006.03.003. Epub 2006 Apr 24. PMID 16632411